CLINICAL TRIAL: NCT00476125
Title: Effects of Dietary Manipulation on Metabolism in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jody Dushay, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007P000017
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Regulation; Fasting; Ketogenic Diet
MeSH Terms: conditions — Fasting | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 day ketogenic diet (Experimental)
  Interventions: Behavioral: Dietary manipulation ketogenic diet
- 12 day ketogenic diet (Experimental)
  Interventions: Behavioral: Dietary Manipulation - 12 day ketogenic diet
- 16 hour fast (Experimental)
  Interventions: Behavioral: 16 Hour Fast

INTERVENTIONS:
Behavioral: Dietary manipulation ketogenic diet — Subjects will consume a ketogenic diet for 3 days.
  Arms: 3 day ketogenic diet
Behavioral: Dietary Manipulation - 12 day ketogenic diet — Subjects will consume a ketogenic diet for 12 days.
  Arms: 12 day ketogenic diet
Behavioral: 16 Hour Fast — Subjects will fast for 16 hours.
  Arms: 16 hour fast

SUMMARY:
This study will examine the potential changes in the blood levels of a recently discovered metabolic regulator in response to changes in diet in healthy adults. Our hypothesis is that in healthy adults key regulatory factors involved in lipid oxidation will respond to changes in diet, particularly fasting and diet-induced ketosis.

DETAILED DESCRIPTION:
There is scant data regarding the metabolic events that occur in humans during ketosis which may be brought about by fasting or ingestion of diets low in carbohydrate.

We aim to employ both fasting and dietary manipulation in order to bring about a ketotic state in healthy human adults. During the study blood levels of key metabolic regulators will be monitored 1) during a 16 hour fast followed by re-feeding and 2) during dietary induction of ketosis followed by re-feeding with a standard meal.

ELIGIBILITY:
Inclusion criteria:

1. Men and women ages 18-60
2. BMI 21-28 kg/m2
3. Stable weight (variation < 3 kg within 6 months of screening visit)
4. Ability to give informed consent
5. Ability to follow verbal and written instructions in English
6. Use of medically approved form of contraception (monophasic oral contraception, intra uterine device, surgical sterilization or 2 combined barrier methods)

Exclusion Criteria:

1. Type 1 or type 2 diabetes mellitus diagnosed according to American Diabetes Association criteria
2. Coronary heart disease (history of myocardial infarction, unstable angina pectoris, or congestive heart failure)
3. Uncontrolled hypertension (BP > 150/90 mmHg on or off antihypertensive medication)
4. Dyslipidemia
5. Tobacco, marijuana or intravenous drug use
6. Shift workers (night shift or alternating day/night shifts)
7. Recent weight loss (> 3 kg within 6 months of the screening visit)
8. Gastroparesis
9. Inflammatory bowel disease
10. Malignancy treated with chemotherapy within the past 3 years
11. History of pancreatitis
12. Depression or psychosis
13. Renal insufficiency (creatinine clearance < 50 ml/min)
14. Transaminases > 2x above the normal range
15. Known liver disease
16. Pregnancy within 6 months of the screening visit
17. Lactation
18. Failure to use medically approved contraceptive methods
19. History of an eating disorder (anorexia, bulimia or laxative abuse)
20. History of surgery for the treatment of obesity (gastric banding, gastric bypass, gastric stapling)
21. New diagnosis of hypo or hyperthyroidism within 1 year of screening visit
22. History of alcohol abuse within the past 5 years
23. Seizure disorder
24. Gout
25. Kidney stones

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Changes in circulating plasma levels of key metabolic regulators | 1 week

SECONDARY OUTCOMES:
A secondary outcome is change in energy expenditure with diet-induced ketosis. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Eleftheria Maratos Flier, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States